CLINICAL TRIAL: NCT06577779
Title: An Open-Label Treatment With Randomization Observation, Investigator-Initiated Study, on the Duration and Efficacy of Jornay PM (Methylphenidate Hydrochloride Extended-Release Capsules) on Adult ADHD Symptoms and Executive Function and Emotional Regulation Throughout the Day Into Early Evening
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01325
Record Dates: First submitted 2024-08-28; First posted 2024-08-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: ADHD; Adult ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Seven weeks of Jornay PM treatment (Active Comparator): Enrolled participants will begin with a two-week observation stabilization before starting treatment with Jornay PM. Participants found to have ≥30% change in their total Adult ADHD Investigator Symptom Rating Scale (AISRS) scores during the two-week observation stabilization period treatment will be discontinued from the study. Remaining participants will initiate a 7 week open-label treatment with Jornay PM.
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsule
- Five weeks of Jornay PM treatment (Experimental): Enrolled participants will begin with a two-week observation stabilization before starting treatment with Jornay PM. Participants found to have ≥30% change in their total Adult ADHD Investigator Symptom Rating Scale (AISRS) scores during the two-week observation stabilization period treatment will be discontinued from the study. Remaining participants will initiate a 5 week open-label treatment with Jornay PM followed by a two week observation period; not receiving Jornay PM.
  Interventions: Drug: Methylphenidate Hydrochloride Extended Release Capsule

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride Extended Release Capsule — Subjects will start at dose of 40mg (DR/ER-MPH) day with titrations of 20mg leading to a maximum dose of 100mg (DR/ER-MPH).
  Other Names: Jornay PM

SUMMARY:
The goal of this study is to extend the efficacy evidence of sustained release methylphenidate compound (JornayPM) in adults with Attention-deficit/hyperactivity disorder (ADHD). JornayPM has recently been approved for treatment of patients 6 years and older with ADHD; the release mechanism is unique among ADHD products in that it is taken in the evening, with effects in the morning upon awakening and then throughout the subsequent day. Of note, to date, there is no clinical data as to the tolerability or clinical effects or dosing in adults with ADHD; therefore the primary aim of this trial is to gather the first set of these data.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-60 years, inclusive at the time of consent
2. Able to provide signed informed consent
3. Any gender
4. Subjects with a current primary Diagnostic and Statistical Manual of Mental Disorders (DSM) -5 diagnosis of ADHD of predominantly inattentive presentation, or combined presentations) as confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) Version 1.2.
5. Subjects who are not receiving any pharmacological treatment for ADHD must have an DSM AISRS 18 item total score of ≥ 28 at screening. Subjects who were previously receiving pharmacological treatment for ADHD at screening must have a minimum total DSM AISRS 18 item score of ≥ 22 at screening
6. Dysthymia and anxiety disorders in remission, but stable on psychiatric medication for three weeks or more at the discretion of principal investigator will be allowed. Medication for these disorders to remain constant for the duration of the protocol.
7. Subjects, who have not used stimulant medication in the past 2 months.
8. Occasional use of marijuana (less than 3 times weekly) will be allowed during screening process until subject is enrolled into the study. After subject is enrolled onto Jornay PM, subject is asked to complete an attestation. The attestation will state that the subject will not consume marijuana while in the study.
9. No illicit substance will be allowed at screening or during the study.

Exclusion Criteria:

1. Known hypersensitivity to methylphenidate, or product components.
2. Concurrent treatment with a monoamine oxidase inhibitor (MAOI), or use of an MAOI within the preceding 14 days.
3. Lifetime bipolar disorder, psychotic disorders, autism, intellectual disability except mood disorders accepted under the inclusion criteria at the discretion of the principal investigator.
4. Active suicidality within past year, or history of suicide attempt in past 2 years
5. Any history of severe past drug dependence determined by the Mini International Neuropsychiatric Interview (MINI) (i.e., a focus of clinical attention or a cause of substantial social or occupational difficulty)
6. Concurrent substance abuse and/or history of substance use within 6 months (except for marijuana use of less than three times a week and/or history of excessive marijuana use of less than three times a week within 6 months).
7. Use of any prescribed benzodiazepine
8. Any unstable medical or neurological condition; clinically significant medical abnormalities such as cardiovascular abnormalities, and any chronic condition of the central nervous system
9. Antidepressants and anti-anxiety agents (including benzodiazepines) taken in stable doses will be allowed, while other psychotropic medications, including hallucinogens, mood stabilizers, antipsychotics will not be allowed
10. Known nonresponse to MPH treatment
11. History of allergic reaction or sensitivity to MPH
12. Female of childbearing age, who are breastfeeding, pregnant, planning to be pregnant or men planning to make a woman pregnant during the study or for one-month post study
13. PI/clinician discretion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Expanded Adult ADHD Investigator Symptom Rating Scale (AISRS) Score from Baseline to Week 3 | Baseline, Week 3
  The expanded AISRS is an 18-item questionnaire assessing symptoms of adult ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate more severe symptoms of ADHD.
Change in Expanded Adult ADHD Investigator Symptom Rating Scale (AISRS) Score from Baseline to Week 10 | Baseline, Week 10
  The expanded AISRS is an 18-item questionnaire assessing symptoms of adult ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate more severe symptoms of ADHD.

SECONDARY OUTCOMES:
Change in Expanded AISRS - Overall Inattentive (IA) Subscale Score | Baseline, Week 3
  9-item subscale of the AISRS assessing inattentive symptoms of ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater overall inattentive symptoms.
Change in Expanded AISRS - Overall Inattentive (IA) Subscale Score | Baseline, Week 10
  9-item subscale of the AISRS assessing inattentive symptoms of ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater overall inattentive symptoms.
Change in Expanded AISRS - Hyperactive/Impulsive (HI) Subscale Score | Baseline, Week 3
  9-item subscale of the AISRS assessing hyperactive/impulsive symptoms of ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater hyperactive/impulsive symptoms.
Change in Expanded AISRS - Hyperactive/Impulsive (HI) Subscale Score | Baseline, Week 10
  9-item subscale of the AISRS assessing hyperactive/impulsive symptoms of ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater hyperactive/impulsive symptoms.
Change from Baseline in Clinical Global Impression-Severity (CGI-S) Scale Score | Baseline, Week 3
  1-item clinician-rated assessment of the severity of a subject's mental illness. The severity of illness is rated as follows: 0 (not assessed), 1 (normal, not at all ill), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most extremely ill subjects). The total score is the numerical ranking provided by the clinician.
Change from Baseline in Clinical Global Impression-Severity (CGI-S) Scale Score | Baseline, Week 10
  1-item clinician-rated assessment of the severity of a subject's mental illness. The severity of illness is rated as follows: 0 (not assessed), 1 (normal, not at all ill), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most extremely ill subjects). The total score is the numerical ranking provided by the clinician.
11-Hours Post-Dose Time-Sensitive ADHD Symptom Scale (TASS) Score at Visit 3 | Week 3 (11-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
11-Hours Post-Dose TASS Score at Visit 4 | Week 4 (11-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
11-Hours Post-Dose TASS Score at Visit 5 | Week 5 (11-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
11-Hours Post-Dose TASS Score at Visit 6 | Week 6 (11-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
11-Hours Post-Dose TASS Score at Visit 7 | Week 7 (11-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
11-Hours Post-Dose TASS Score at Visit 8 | Week 8 (11-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
11-Hours Post-Dose TASS Score at Visit 9 | Week 9 (11-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
11-Hours Post-Dose TASS Score at Visit 10 | Week 10 (11-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
16-Hours Post-Dose TASS Score at Visit 3 | Week 3 (16-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
16-Hours Post-Dose TASS Score at Visit 4 | Week 4 (16-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
16-Hours Post-Dose TASS Score at Visit 5 | Week 5 (16-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
16-Hours Post-Dose TASS Score at Visit 6 | Week 6 (16-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
16-Hours Post-Dose TASS Score at Visit 7 | Week 7 (16-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
16-Hours Post-Dose TASS Score at Visit 8 | Week 8 (16-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
16-Hours Post-Dose TASS Score at Visit 9 | Week 9 (16-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
16-Hours Post-Dose TASS Score at Visit 10 | Week 10 (16-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
21-Hours Post-Dose TASS Score at Visit 3 | Week 3 (21-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
21-Hours Post-Dose TASS Score at Visit 4 | Week 4 (21-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
21-Hours Post-Dose TASS Score at Visit 5 | Week 5 (21-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
21-Hours Post-Dose TASS Score at Visit 6 | Week 6 (21-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
21-Hours Post-Dose TASS Score at Visit 7 | Week 7 (21-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
21-Hours Post-Dose TASS Score at Visit 8 | Week 8 (21-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
21-Hours Post-Dose TASS Score at Visit 9 | Week 9 (21-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
21-Hours Post-Dose TASS Score at Visit 10 | Week 10 (21-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
24-Hours Post-Dose TASS Score at Visit 3 | Week 3 (24-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
24-Hours Post-Dose TASS Score at Visit 4 | Week 4 (24-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
24-Hours Post-Dose TASS Score at Visit 5 | Week 5 (24-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
24-Hours Post-Dose TASS Score at Visit 6 | Week 6 (24-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
24-Hours Post-Dose TASS Score at Visit 7 | Week 7 (24-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
24-Hours Post-Dose TASS Score at Visit 8 | Week 8 (24-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
24-Hours Post-Dose TASS Score at Visit 9 | Week 9 (24-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
24-Hours Post-Dose TASS Score at Visit 10 | Week 10 (24-hours Post-Dose)
  18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
11-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 3 | Week 3 (11-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
11-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 8 | Week 8 (11-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
11-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 10 | Week 10 (11-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
16-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 3 | Week 3 (16-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
16-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 8 | Week 8 (16-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
16-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 10 | Week 10 (16-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
21-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 3 | Week 3 (21-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
21-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 8 | Week 8 (21-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
21-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 10 | Week 10 (21-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
24-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 3 | Week 3 (24-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
24-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 8 | Week 8 (24-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
24-Hours Post-Dose Smoothness of Effect Scale (AMSES) Score at Visit 10 | Week 10 (24-hours Post-Dose)
  5-item assessment of the smoothness of effect of ADHD medication throughout the day following dosing. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 20; higher scores indicate greater smoothness of effect of medication.
Change in Adult ADHD Self Report Scale (ASRS) Symptom Checklist Score | Baseline, Week 3
  The ASRS is a 31-item questionnaire assessing frequency of ADHD symptoms over the previous 7 days. Items are rate on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 124; higher scores indicate greater frequency of ADHD symptoms.
Change in Adult ADHD Self Report Scale (ASRS) Symptom Checklist Score | Baseline, Week 10
  The ASRS is a 31-item questionnaire assessing frequency of ADHD symptoms over the previous 7 days. Items are rate on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0 to 124; higher scores indicate greater frequency of ADHD symptoms.
Change in Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) Score | Baseline, Week 3
  The BRIEF-A is a 75-item self-report questionnaire assessing behavioral issues. Items are rated on a 3-point Likert scale: 0 (never), 1 (sometimes), and 2 (often).
Change in Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) Score | Baseline, Week 10
  The BRIEF-A is a 75-item self-report questionnaire assessing behavioral issues. Items are rated on a 3-point Likert scale: 0 (never), 1 (sometimes), and 2 (often).

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Adler, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The summary data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Terry.Leon@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.